CLINICAL TRIAL: NCT03666143
Title: A Phase 1b Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of Sitravatinib in Combination With Tislelizumab in Patients With Advanced Solid Tumors
Brief Title: A Phase 1b Study to Assess Sitravatinib in Combination With Tislelizumab in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-900-103; CTR20181404 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2018-08-21; First posted 2018-09-11 (Actual); Results first posted 2024-06-17 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — sitravatinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sitravatinib + Tislelizumab (Experimental): Sitravatinib 120 mg was administered orally once daily in combination with tislelizumab 200 mg intravenously (IV) once every 3 weeks
  Interventions: Drug: Sitravatinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: Sitravatinib — Administered orally as a capsule
  Other Names: MGCD516
Drug: Tislelizumab — Administered intravenously
  Other Names: BGB-A317; Tevimbra

SUMMARY:
This was an open-label, multicenter, non-randomized Phase 1b clinical trial for participants with histologically or cytologically confirmed locally advanced or metastatic tumors including non-squamous or squamous non-small cell lung cancer (NSCLC), renal cell carcinoma (RCC), ovarian cancer (OC), or melanoma.

DETAILED DESCRIPTION:
All participants received sitravatinib 120 mg orally once daily in combination with tislelizumab 200 mg intravenously (IV) once every 3 weeks until occurrence of progressive disease, unacceptable toxicity, death, withdrawal of consent, or study termination by sponsor. Participants were enrolled according to their tumor type and prior anti-programmed cell death protein-1 (PD-1)/PD-L1 antibody treatment into the following cohorts:

* Cohort A: Anti-PD-1/PD-L1 antibody refractory/resistant metastatic, non-squamous NSCLC
* Cohort B: Anti-PD-1/PD-L1 antibody naïve metastatic, non-squamous NSCLC
* Cohort C: Anti-PD-1/PD-L1 antibody refractory/resistant metastatic or advanced RCC
* Cohort D: Metastatic or advanced RCC without prior systemic therapy
* Cohort E: Anti-PD-1/PD-L1 antibody naïve recurrent and platinum resistant epithelial OC
* Cohort F: Anti-PD-1/PD-L1 antibody treated metastatic, squamous NSCLC
* Cohort G: Anti-PD-1/PD-L1 antibody refractory/resistant unresectable or metastatic melanoma
* Cohort H: PD-L1 positive, locally advanced or metastatic, non-squamous NSCLC without prior systemic treatment in the metastatic setting
* Cohort I: PD-L1 positive, locally advanced or metastatic, squamous NSCLC without prior systemic treatment in the metastatic setting

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the Schedule of Assessments
2. Age ≥ 18 years on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place)
3. At least 1 measurable lesion as defined by RECIST v1.1
4. Provide archival tumor tissue (formalin-fixed paraffin-embedded block [FFPE] with tumor tissue or unstained slides), if available.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
6. Adequate hematologic and end-organ function
7. Participants with inactive/asymptomatic carrier, chronic, or active hepatitis B virus (HBV) must have HBV deoxyribonucleic acid (DNA) < 500 IU/mL (or 2500 copies/mL) at Screening
8. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and ≥ 120 days after the last dose of study drugs and have a negative serum pregnancy test ≤ 7 days of first dose of study drugs
9. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥ 120 days after the last dose of study drugs

Exclusion Criteria:

1. Unacceptable toxicity on prior anti-PD-1/PD-L1 treatment
2. Active leptomeningeal disease or uncontrolled brain metastasis
3. Active autoimmune diseases or history of autoimmune diseases that may relapse
4. Any active malignancy ≤ 2 years
5. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before first dose of study drugs
6. History of interstitial lung disease, noninfectious pneumonitis or uncontrolled diseases, including pulmonary fibrosis, acute lung diseases, etc.
7. Severe chronic or active infections (including tuberculosis infection, etc.) requiring systemic antibacterial, antifungal or antiviral therapy, within 14 days prior to first dose of study drugs
8. Known history of human immunodeficiency virus (HIV) infection
9. Participants with active hepatitis C infection
10. Any major surgical procedure requiring general anesthesia ≤ 28 days before first dose of study drugs
11. Prior allogeneic stem cell transplantation or organ transplantation
12. Hypersensitivity to tislelizumab or sitravatinib, to any ingredient in the formulation, or to any component of the container
13. Bleeding or thrombotic disorders or use of anticoagulants such as warfarin or similar agents requiring therapeutic international normalized ratio (INR) monitoring within 6 months before first dose of study drugs
14. Concurrent participation in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (19):
- Australia (6):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Icon Cancer Foundation, South Brisbane, Queensland
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Nucleus Network, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- China (13):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Guo J, Zhou Q, Huang D, Yu X, Zhao J, Chu Q, Ma Z, Millward M, Gao B, Goh J, Markman B, Voskoboynik M, Gan H, Coward J, Chen C, Xiang X, Qui J, Xu Y, Yang L, Wu YL. A phase 1b study to assess safety, tolerability, pharmacokinetics, and preliminary antitumor activity of sitravatinib in combination with tislelizumab in patients (pts) with advanced solid tumors. Chinese Society of Clinical Oncology. 2019.
- [Background] Zhao J, Yu X, Huang D, Ma Z, Gao B, Cui J, Chu Q, Zhou Q, Sun M, Day D, Wu J, Pan H, Wang L, Voskoboynik M, Wang Z, Liu Y, Li H, Zhang J, Peng Y, Wu YL. SAFFRON-103: a phase 1b study of the safety and efficacy of sitravatinib combined with tislelizumab in patients with locally advanced or metastatic non-small cell lung cancer. J Immunother Cancer. 2023 Feb;11(2):e006055. doi: 10.1136/jitc-2022-006055. PMID 36808075
- [Derived] Wang X, Pan H, Cui J, Chen X, Yoon WH, Carlino MS, Li X, Li H, Zhang J, Sun J, Guo J, Cui C. SAFFRON-103: a phase Ib study of sitravatinib plus tislelizumab in anti-PD-(L)1 refractory/resistant advanced melanoma. Immunotherapy. 2024 Mar;16(4):243-256. doi: 10.2217/imt-2023-0130. Epub 2024 Jan 10. PMID 38197138

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants across study centers in Australia and China.
Period: Overall Study
Arm/Group | Sitravatinib + Tislelizumab
Started | 216
Completed | 0
Not Completed | 216
Not completed — Death | 158
Not completed — Sponsor Decision | 31
Not completed — Withdrawal by Subject | 11
Not completed — Lost to Follow-up | 5
Not completed — Physician Decision | 1
Not completed — Rolled into extension study | 9
Not completed — Progressive Disease | 1

BASELINE CHARACTERISTICS:
Groups:
- Sitravatinib + Tislelizumab: Sitravatinib 120 mg was administered orally once daily in combination with tislelizumab 200 mg IV once every 3 weeks
Arm/Group | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 216
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.2 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 213
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 143
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 70
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with treatment-emergent AEs (TEAEs) and serious adverse events (SAEs), which includes laboratory tests, physical exams, electrocardiogram results and vital signs; TEAE was defined as an adverse event that had an onset date or a worsening in severity from baseline (pretreatment) on or after the first dose of study drug(s) up to 30 days following last dose of study drug(s) or initiation of a new anticancer therapy, whichever occurs first.
Time Frame: Up to approximately 4 years and 2 months
Population: The Safety Analysis Set is defined as all participants who received at least 1 dose of any study drug (any component of the combination therapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 216
Participants
  At least 1 TEAE | 216
  At least 1 SAE | 120

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with confirmed complete response (CR) or partial response (PR) as determined by the investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Efficacy was evaluated by cohort, as pre-specified in the statistical analysis plan.
Time Frame: Up to approximately 4 years and 2 months
Population: The Efficacy Evaluable Analysis Set consists of all treated participants in the Safety Analysis Set with measurable baseline assessment per RECIST 1.1 who had at least one evaluable post-baseline tumor assessment unless treatment was discontinued due to clinical disease progression or early death (within 13 weeks of the first dose date)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Sitravatinib + Tislelizumab: Sitravatinib 120 mg was administered orally once daily in combination with tislelizumab 200 mg IV once every 3 weeks. Dose regimen was investigated in the following cohorts:
  * Cohort A: Anti-PD-1/PD-L1 antibody refractory/resistant (R/R) metastatic non-squamous non-small cell lung cancer (NSCLC)
  * Cohort B: Anti-PD-1/PD-L1 antibody naïve metastatic non-squamous NSCLC
  * Cohort C: Anti-PD-1/PD-L1 antibody R/R metastatic or advanced renal cell carcinoma (RCC)
  * Cohort D: Metastatic or advanced RCC without prior systemic therapy
  * Cohort E: Anti-PD-1/PD-L1 antibody naïve recurrent and platinum-resistant epithelial ovarian cancer (OC)
  * Cohort F: Anti-PD-1/PD-L1 antibody treated metastatic squamous NSCLC
  * Cohort G: Anti-PD-1/PD-L1 antibody R/R unresectable or metastatic melanoma
  * Cohort H: PD-L1 positive locally advanced or metastatic non-squamous NSCLC without prior systemic treatment in the metastatic setting
  * Cohort I: PD-L1 positive locally advanced or metastatic squamous NSCLC without prior systemic treatment in the metastatic setting
Arm/Group | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 199
Percentage of participants
  Cohort A: NSCLC: number analyzed (Participants) | 23
  Cohort A: NSCLC | 4.3 [0.1 to 21.9]
  Cohort B: NSCLC: number analyzed (Participants) | 21
  Cohort B: NSCLC | 23.8 [8.2 to 47.2]
  Cohort C: RCC: number analyzed (Participants) | 3
  Cohort C: RCC | 66.7 [9.4 to 99.2]
  Cohort D: RCC: number analyzed (Participants) | 3
  Cohort D: RCC | 0.0 [0.0 to 70.8]
  Cohort E: OC: number analyzed (Participants) | 59
  Cohort E: OC | 28.8 [17.8 to 42.1]
  Cohort F: NSCLC: number analyzed (Participants) | 22
  Cohort F: NSCLC | 18.2 [5.2 to 40.3]
  Cohort G: Melanoma: number analyzed (Participants) | 25
  Cohort G: Melanoma | 36.0 [18.0 to 57.5]
  Cohort H: NSCLC: number analyzed (Participants) | 20
  Cohort H: NSCLC | 60.0 [36.1 to 80.9]
  Cohort I: NSCLC: number analyzed (Participants) | 23
  Cohort I: NSCLC | 30.4 [13.2 to 52.9]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the first determination of an objective response until the first documentation of progressive disease, whichever comes first, as assessed by the investigator using RECIST v1.1. Results are reported for cohorts with responders, defined as CR or PR. Efficacy was evaluated by cohort, as pre-specified in the statistical analysis plan.
Time Frame: Up to approximately 4 years and 2 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Sitravatinib + Tislelizumab: Sitravatinib 120 mg was administered orally once daily in combination with tislelizumab 200 mg IV once every 3 weeks. Dose regimen was investigated in the following cohorts:
  * Cohort A: Anti-PD-1/PD-L1 antibody R/R metastatic non-squamous NSCLC
  * Cohort B: Anti-PD-1/PD-L1 antibody naïve metastatic non-squamous NSCLC
  * Cohort C: Anti-PD-1/PD-L1 antibody R/R metastatic or advanced RCC
  * Cohort E: Anti-PD-1/PD-L1 antibody naïve recurrent and platinum-resistant epithelial OC
  * Cohort F: Anti-PD-1/PD-L1 antibody treated metastatic squamous NSCLC
  * Cohort G: Anti-PD-1/PD-L1 antibody R/R unresectable or metastatic melanoma
  * Cohort H: PD-L1 positive locally advanced or metastatic non-squamous NSCLC without prior systemic treatment in the metastatic setting
  * Cohort I: PD-L1 positive locally advanced or metastatic squamous NSCLC without prior systemic treatment in the metastatic setting
Arm/Group | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 57
Months
  Cohort A: NSCLC: number analyzed (Participants) | 1
  Cohort A: NSCLC | 3.1 [NA to NA] — NA = Data not estimable due to low number of participants with events
  Cohort B: NSCLC: number analyzed (Participants) | 5
  Cohort B: NSCLC | 17.9 [2.9 to NA] — NA = Data not estimable due to low number of participants with events
  Cohort C: RCC: number analyzed (Participants) | 2
  Cohort C: RCC | 11.4 [9.7 to NA] — NA = Data not estimable due to low number of participants with events
  Cohort E: OC: number analyzed (Participants) | 17
  Cohort E: OC | 5.6 [2.8 to 12.5]
  Cohort F: NSCLC: number analyzed (Participants) | 4
  Cohort F: NSCLC | 6.9 [3.4 to NA] — NA = Data not estimable due to low number of participants with events
  Cohort G: Melanoma: number analyzed (Participants) | 9
  Cohort G: Melanoma | 19.1 [2.8 to NA] — NA = Data not estimable due to low number of participants with events
  Cohort H: NSCLC: number analyzed (Participants) | 12
  Cohort H: NSCLC | 9.7 [5.6 to 15.9]
  Cohort I: NSCLC: number analyzed (Participants) | 7
  Cohort I: NSCLC | 8.1 [5.5 to NA] — NA = Data not estimable due to low number of participants with events

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with best overall response as CR, PR, or stable disease (SD) as assessed by the investigator using RECIST v1.1. Efficacy was evaluated by cohort, as pre-specified in the statistical analysis plan.
Time Frame: Up to approximately 4 years and 2 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Sitravatinib + Tislelizumab: Sitravatinib 120 mg was administered orally once daily in combination with tislelizumab 200 mg IV once every 3 weeks. Dose regimen was investigated in the following cohorts:
  * Cohort A: Anti-PD-1/PD-L1 antibody R/R metastatic non-squamous NSCLC
  * Cohort B: Anti-PD-1/PD-L1 antibody naïve metastatic non-squamous NSCLC
  * Cohort C: Anti-PD-1/PD-L1 antibody R/R metastatic or advanced RCC
  * Cohort D: Metastatic or advanced RCC without prior systemic therapy
  * Cohort E: Anti-PD-1/PD-L1 antibody naïve recurrent and platinum-resistant epithelial OC
  * Cohort F: Anti-PD-1/PD-L1 antibody treated metastatic squamous NSCLC
  * Cohort G: Anti-PD-1/PD-L1 antibody R/R unresectable or metastatic melanoma
  * Cohort H: PD-L1 positive locally advanced or metastatic non-squamous NSCLC without prior systemic treatment in the metastatic setting
  * Cohort I: PD-L1 positive locally advanced or metastatic squamous NSCLC without prior systemic treatment in the metastatic setting
Arm/Group | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 199
Percentage of participants
  Cohort A: NSCLC: number analyzed (Participants) | 23
  Cohort A: NSCLC | 78.3 [56.3 to 92.5]
  Cohort B: NSCLC: number analyzed (Participants) | 21
  Cohort B: NSCLC | 85.7 [63.7 to 97.0]
  Cohort C: RCC: number analyzed (Participants) | 3
  Cohort C: RCC | 100.0 [29.2 to 100.0]
  Cohort D: RCC: number analyzed (Participants) | 3
  Cohort D: RCC | 100.0 [29.2 to 100.0]
  Cohort E: OC: number analyzed (Participants) | 59
  Cohort E: OC | 79.7 [67.2 to 89.0]
  Cohort F: NSCLC: number analyzed (Participants) | 22
  Cohort F: NSCLC | 90.9 [70.8 to 98.9]
  Cohort G: Melanoma: number analyzed (Participants) | 25
  Cohort G: Melanoma | 88.0 [68.8 to 97.5]
  Cohort H: NSCLC: number analyzed (Participants) | 20
  Cohort H: NSCLC | 85.0 [62.1 to 96.8]
  Cohort I: NSCLC: number analyzed (Participants) | 23
  Cohort I: NSCLC | 78.3 [56.3 to 92.5]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from the date of first dose to the date of first documentation of progressive disease or death, whichever comes first, as assessed by the investigator using RECIST v1.1. Efficacy was evaluated by cohort, as pre-specified in the statistical analysis plan.
Time Frame: Up to approximately 4 years and 2 months
Population: The Safety Analysis Set for this endpoint is defined as all participants who received at least 1 dose of any study drug (any component of the combination therapy) and who met tumor type criteria per latest protocol amendment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 209
Months
  Cohort A: NSCLC: number analyzed (Participants) | 24
  Cohort A: NSCLC | 4.2 [2.7 to 5.8]
  Cohort B: NSCLC: number analyzed (Participants) | 22
  Cohort B: NSCLC | 7.0 [2.7 to 11.2]
  Cohort C: RCC: number analyzed (Participants) | 3
  Cohort C: RCC | 15.9 [11.1 to NA] — NA = Data not estimable due to low number of participants with events
  Cohort D: RCC: number analyzed (Participants) | 3
  Cohort D: RCC | 2.7 [2.6 to NA] — NA = Data not estimable due to low number of participants with events
  Cohort E: OC: number analyzed (Participants) | 63
  Cohort E: OC | 4.1 [3.5 to 5.1]
  Cohort F: NSCLC: number analyzed (Participants) | 23
  Cohort F: NSCLC | 5.3 [4.1 to 8.2]
  Cohort G: Melanoma: number analyzed (Participants) | 25
  Cohort G: Melanoma | 6.7 [4.1 to 29.7]
  Cohort H: NSCLC: number analyzed (Participants) | 22
  Cohort H: NSCLC | 10.9 [5.1 to 15.3]
  Cohort I: NSCLC: number analyzed (Participants) | 24
  Cohort I: NSCLC | 5.4 [2.8 to 9.5]

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Sitravatinib
Time Frame: Predose and up to 24 hours post dose on Cycle 1 Day 1 (C1D1) and Cycle 1 Day 21 (C1D21); 21 days per cycle
Population: The Sitravatinib Pharmacokinetic (PK) Analysis Set includes all participants who contributed at least 1 quantifiable PK sample for sitravatinib
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 42
nanograms/milliliter (ng/mL)
  C1D1 | 49.49 (82.688)
  C1D21: number analyzed (Participants) | 27
  C1D21 | 98.36 (68.908)

7. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for Sitravatinib
Time Frame: Predose and up to 24 hours post dose on C1D1 and C1D21; 21 days per cycle
Population: The Sitravatinib PK Analysis Set includes all participants who contributed at least 1 quantifiable PK sample for sitravatinib
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 42
Hours (h)
  C1D1 | 6.09 [2.0 to 24.8]
  C1D21: number analyzed (Participants) | 27
  C1D21 | 6.08 [0.0 to 23.2]

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Time Point (AUC(0-t)) for Sitravatinib
Time Frame: Predose and up to 24 hours post dose on C1D1 and C1D21; 21 days per cycle
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 42
h*ng/mL
  C1D1 | 414.01 (115.833)
  C1D21: number analyzed (Participants) | 27
  C1D21 | 1539.96 (83.010)

9. Secondary Outcome: Clearance After Oral Administration (CL/F) for Sitravatinib
Time Frame: Predose and up to 24 hours post dose on C1D1 and C1D21; 21 days per cycle
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 14
Liters/hour
  C1D1: number analyzed (Participants) | 7
  C1D1 | 72.89 (148.368)
  C1D21 | 58.30 (58.470)

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve During the Dosing Interval (AUC(0-tau)) for Sitravatinib
Time Frame: Predose and up to 24 hours post dose on C1D1 and C1D21; 21 days per cycle
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 14
h*ng/mL
  C1D1: number analyzed (Participants) | 10
  C1D1 | 1050.57 (75.432)
  C1D21 | 2058.23 (58.470)

11. Secondary Outcome: Observed Accumulation Ratio (Ro) for AUC0-tau for Sitravatinib
Description: Presented as geometric mean ratio and confidence interval, transformed from the difference of least square means and confidence interval of the least square differences in the logarithmic scale by exponentiation
Time Frame: Predose and up to 24 hours post dose on C1D1 and C1D21; 21 days per cycle
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 7
Ratio | 1.83 [1.18 to 2.82]

12. Secondary Outcome: Observed Accumulation Ratio (Ro) for Cmax for Sitravatinib
Description: as for outcome 11
Time Frame: Predose and up to 24 hours post dose on C1D1 and C1D21; 21 days per cycle
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 27
Ratio | 2.23 [1.69 to 2.95]

ADVERSE EVENTS:
Time Frame: From the first dose up to 30 days after the last dose of study drug; Up to approximately 4 years and 2 months
Description: An adverse event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study drug, whether considered related to study drug or not.
Arm/Group | Sitravatinib + Tislelizumab
All-Cause Mortality (participants affected / at risk) | 158/216
Serious Adverse Events (participants affected / at risk) | 120/216
Other Adverse Events (participants affected / at risk) | 213/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitravatinib + Tislelizumab (N=216)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2)
Immune-mediated myocarditis (Cardiac disorders) | 2 (2)
Myocarditis (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Adrenocortical insufficiency acute (Endocrine disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypophysitis (Endocrine disorders) | 1 (1)
Immune-mediated hyperthyroidism (Endocrine disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 4 (6)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (12)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 4 (8)
Large intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 6 (12)
Terminal ileitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7)
Death (General disorders) | 9 (9)
Device related thrombosis (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 8 (8)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (4)
Hepatic pain (Hepatobiliary disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (2)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 3 (3)
Appendicitis perforated (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Furuncle (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (3)
Pneumonia (Infections and infestations) | 10 (11)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4)
Urosepsis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Incarcerated parastomal hernia (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 2 (2)
Transaminases increased (Investigations) | 3 (3)
Troponin I increased (Investigations) | 2 (2)
Troponin increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Device occlusion (Product Issues) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Aortic dissection (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Jugular vein thrombosis (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitravatinib + Tislelizumab (N=216)
Anaemia (Blood and lymphatic system disorders) | 39 (56)
Sinus bradycardia (Cardiac disorders) | 7 (7)
Sinus tachycardia (Cardiac disorders) | 8 (12)
Ventricular extrasystoles (Cardiac disorders) | 7 (10)
Hyperthyroidism (Endocrine disorders) | 15 (17)
Hypothyroidism (Endocrine disorders) | 71 (78)
Abdominal distension (Gastrointestinal disorders) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 30 (39)
Abdominal pain upper (Gastrointestinal disorders) | 25 (28)
Constipation (Gastrointestinal disorders) | 46 (52)
Diarrhoea (Gastrointestinal disorders) | 114 (224)
Dry mouth (Gastrointestinal disorders) | 14 (14)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 (16)
Mouth ulceration (Gastrointestinal disorders) | 19 (22)
Nausea (Gastrointestinal disorders) | 67 (86)
Stomatitis (Gastrointestinal disorders) | 24 (28)
Toothache (Gastrointestinal disorders) | 10 (11)
Vomiting (Gastrointestinal disorders) | 57 (97)
Asthenia (General disorders) | 8 (9)
Fatigue (General disorders) | 45 (52)
Influenza like illness (General disorders) | 10 (10)
Malaise (General disorders) | 16 (17)
Non-cardiac chest pain (General disorders) | 7 (7)
Oedema peripheral (General disorders) | 12 (12)
Pyrexia (General disorders) | 25 (39)
Hepatic function abnormal (Hepatobiliary disorders) | 8 (17)
Pneumonia (Infections and infestations) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 8 (9)
Urinary tract infection (Infections and infestations) | 21 (27)
Alanine aminotransferase increased (Investigations) | 101 (198)
Aspartate aminotransferase increased (Investigations) | 97 (181)
Bilirubin conjugated increased (Investigations) | 22 (35)
Blood alkaline phosphatase increased (Investigations) | 19 (27)
Blood bilirubin increased (Investigations) | 21 (38)
Blood cholesterol increased (Investigations) | 24 (51)
Blood creatine phosphokinase MB increased (Investigations) | 26 (42)
Blood creatine phosphokinase increased (Investigations) | 43 (95)
Blood creatinine increased (Investigations) | 13 (20)
Blood lactate dehydrogenase increased (Investigations) | 33 (55)
Blood potassium decreased (Investigations) | 7 (23)
Blood pressure increased (Investigations) | 15 (22)
Blood thyroid stimulating hormone increased (Investigations) | 26 (33)
Electrocardiogram QT prolonged (Investigations) | 14 (14)
Electrocardiogram T wave abnormal (Investigations) | 13 (40)
Gamma-glutamyltransferase increased (Investigations) | 28 (51)
Neutrophil count decreased (Investigations) | 11 (16)
Neutrophil count increased (Investigations) | 7 (13)
Platelet count decreased (Investigations) | 23 (44)
Urobilinogen urine increased (Investigations) | 9 (14)
Weight decreased (Investigations) | 82 (98)
Weight increased (Investigations) | 7 (8)
White blood cell count decreased (Investigations) | 14 (23)
White blood cell count increased (Investigations) | 7 (14)
White blood cells urine positive (Investigations) | 11 (32)
Decreased appetite (Metabolism and nutrition disorders) | 71 (77)
Hyperglycaemia (Metabolism and nutrition disorders) | 21 (40)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 19 (47)
Hyperuricaemia (Metabolism and nutrition disorders) | 16 (34)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 47 (63)
Hypocalcaemia (Metabolism and nutrition disorders) | 26 (47)
Hypochloraemia (Metabolism and nutrition disorders) | 7 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 30 (75)
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 (23)
Hyponatraemia (Metabolism and nutrition disorders) | 29 (43)
Hypophosphataemia (Metabolism and nutrition disorders) | 14 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (26)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (12)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (12)
Dizziness (Nervous system disorders) | 18 (19)
Headache (Nervous system disorders) | 26 (32)
Hypoaesthesia (Nervous system disorders) | 7 (7)
Lethargy (Nervous system disorders) | 8 (8)
Insomnia (Psychiatric disorders) | 14 (14)
Proteinuria (Renal and urinary disorders) | 41 (76)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (30)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 35 (36)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 (22)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 (15)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 63 (83)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (12)
Rash (Skin and subcutaneous tissue disorders) | 38 (49)
Hypertension (Vascular disorders) | 81 (97)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT03666143/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT03666143/SAP_001.pdf